CLINICAL TRIAL: NCT04677348
Title: Comparison of Analgesic Effect of Pericapsular Nerve Group Block and Suprainguinal Fascia Iliaca Compartment Block on Dynamic Pain in Patients Undergoing Hip Fracture Surgery: a Randomized Controlled Trial
Brief Title: Comparison of PENG Block and FICB in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-1822
Record Dates: First submitted 2020-12-10; First posted 2020-12-21 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Hip Fractures; Regional Anesthesia
Keywords: pericapsular nerve group block; fascia iliaca compartment block; hip fracture; regional anesthesia; dynamic pain
MeSH Terms: conditions — Hip Fractures | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Experimental): pericapsular nerve group (PENG) block before surgery
  Interventions: Procedure: Pericapsular nerve group (PENG) block
- FICB group (Active Comparator): suprainguinal fascia iliaca compartment block (FICB) before surgery
  Interventions: Procedure: Fascia iliaca compartment block (FICB)

INTERVENTIONS:
Procedure: Pericapsular nerve group (PENG) block — ultrasound-guided PENG block with 0.3% ropivacaine 20cc
  Arms: PENG group
Procedure: Fascia iliaca compartment block (FICB) — ultrasound-guided suprainguinal FICB with 0.3% ropivacaine 30cc
  Arms: FICB group

SUMMARY:
Fascia iliaca compartment block (FICB) has been considered the block of choice for patients with hip fracture. However, pericapsular nerve group (PENG) block, one of the relatively newly-developed blocks, could be also used for analgesia in patients with hip fracture. Since PENG block could block the accessory obturator nerve, PENG block might have greater analgesic effects compared to FICB theoretically. However, the comparison of these two blocks in patients with hip fracture has not performed in clinical setting. Thus, we aimed to compare the analgesic effect of PENG block and FICB.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-4
* age: ≥19
* baseline pain score (associated with hip fracture): ≥4

Exclusion Criteria:

* patients who do not agree to participate in this study
* patients with uncontrolled hypertension, hyperthyroidism, severe dementia
* allergic to ropivacaine
* contraindicated to spinal anesthesia due to coagulopathy, severe aortic stenosis/mitral stenosis, or active infection on lumbar region
* patients who are considered ineligible with any other reason by investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of each block (Pain score) | before surgery
  We will assess the dynamic pain (pain during a movement) using NRS before and 20-30min after applying the assigned block. Then, we will calculate the change of NRS at the two time-points.
  NRS: Numerical rating scale (0, no pain; 10, the worst pain imaginable)

SECONDARY OUTCOMES:
change of blood pressure (systolic, diastolic, mean blood pressure) | before surgery
  We will evaluate the blood pressure before and 20-30min after applying the assigned block. Then, we will calculate the change of blood pressure at the two time-points.
postoperative pain score | postoperative 6, 24, 48hours
  resting and dynamic pain using NRS at postoperative 6, 24, 48hours
  NRS: Numerical rating scale (0, no pain; 10, the worst pain imaginable)
postoperative opioid consumption | postoperative 24, 48hours
  morphine-equivalent dose
postoperative motor function | postoperative 6, 24, 48hours
  motor function of quadriceps femoris
  grade5: normal power grade4: movement possible against some resistance grade3: movement against gravity but not resistance grade2: movement possible if gravity eliminated grade1: flicker of contraction possible grade0: complete paralysis
change of heart rate | before surgery
  We will evaluate the heart rate before and 20-30 min after applying the assigned block. Then, we will calculate the change of heart rate at the two time-points.

CONTACTS AND LOCATIONS:
Overall Officials: Won Uk Koh, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koh WU, Kim H, Kim YJ, Park JI, Yeo HJ, Ro YJ, Kim HJ. Comparison of analgesic effect of pericapsular nerve group block and supra-inguinal fascia iliaca compartment block on dynamic pain in patients with hip fractures: a randomized controlled trial. Reg Anesth Pain Med. 2025 Aug 5;50(8):635-640. doi: 10.1136/rapm-2024-105627. PMID 38866559